CLINICAL TRIAL: NCT03486106
Title: Music Distraction and Its Influence on Anesthetic Requirements During Elective Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20010566
Record Dates: First submitted 2018-03-20; First posted 2018-04-03 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia; Functional; Surgery
MeSH Terms: interventions — Music Therapy; Propofol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Headphones without music (Placebo Comparator): Participants in the control group will receive noise-cancelling wireless headphones that will not play any noise throughout the procedure. They will also receive propofol for sedation as needed.
  Interventions: Other: Headphones; Drug: Propofol
- Headphones with music (Experimental): Participants in the experimental group will receive the same noise-cancelling wireless headphones but will be permitted to listen to the music of their choice while in the operating room. They will also receive propofol for sedation as needed.
  Interventions: Other: Music; Other: Headphones; Drug: Propofol

INTERVENTIONS:
Other: Music — Music will be provided via Spotify, which is an Internet streaming music service, and will be played through headphones; this way, no other individual in the operating room will be distracted or influenced by the patient's music selection.
  Arms: Headphones with music
Other: Headphones — All participants will receive noise-cancelling wireless headphones that they will wear in the operating room during the procedure.
Drug: Propofol — All participants will receive intravenous doses of propofol; the timing and frequency of the doses will be given when the patient indicates (by squeezing a rubber duckie) that he/she wants sedation medication.

SUMMARY:
This study evaluates the effect of music and its influence on anesthetic requirements during total knee replacement surgery. Half of the participants will receive noise-cancelling headphones in the operating room, and the other half of participants will receive noise-cancelling headphones with music playing.

DETAILED DESCRIPTION:
Prior to surgery, patient participants will receive a combined spinal-epidural per VCU total joint protocol; the following steps are considered standard of care and not considered study procedures. The combined spinal-epidural procedure creates complete numbness below the abdomen down to the feet, which negates the need for general anesthesia. For patient comfort during the combined-spinal epidural procedure, a one-time dose of 2 milligrams of intravenous midazolam will be given; this dose is adequate for reducing anxiety while allowing the patient to maintain conversation with health care providers if necessary. The standard intrathecal dose for total knee replacement at our institution is 15 mg bupivacaine and 0.2 mg preservative-free morphine; this dose will provide complete numbness to the lower extremities for approximately 3-6 hours. After this dose is administered, the patient will then be positioned appropriately in the operating room and vital signs will monitored per standard protocol.

Each patient participant will be randomized to one of two groups. Participants in the control group will receive noise-cancelling wireless headphones that will not play any noise throughout the procedure. Participants in the experimental group will receive the same noise-cancelling wireless headphones but will be permitted to listen to the music of their choice while in the operating room. Music will be provided via Spotify, which is an Internet streaming music service, and will be played through headphones; this way, no other individual in the operating room will be distracted or influenced by the patient's music selection. Participants will not be able to change the Spotify channel. We will be using the paid Spotify service with no commercials. If participants opt to have the music stopped, we will withdraw them from the study and continue standard of care. The participants will have the music playing for about two hours. If the participant has no music preference, the music will be chosen for them and it will be the same for all participants that have no preference. The volume will be adjusted in the operating room until the participant approves of the volume by saying "yes, the volume is good" or giving another verbal cue of approval.The music will continue playing until the surgical procedure is complete and the patient has reached the post-anesthesia recovery unit.

As stated previously, spinal anesthesia provides numbness that negates the need for general anesthesia, but patients often times need additional sedation, which will be defined as anesthesia medication that is used to treat patient anxiety and discomfort in the operating room. Patient participants in both groups will receive sedation via the same protocol, which is outlined below.

Sedation will only be given as needed per patient request; the patient will be given a noise-making device (such as a rubber duckie that makes sound when squeezed) that will inform the anesthesia provider that the patient is uncomfortable and needs some sedation. A weight based dose of 0.3 micrograms per kilogram of intravenous propofol will be given for each patient request. This dose is expected to provide amnesia or light sleep for a few minutes. For patient safety, if the patient requests sedation more than once within a two minute window, the anesthesia provider will not administer any more medication during this two minute period. Additionally, the anesthesia provider may withhold sedation if he or she determines with physical exam and hemodynamic monitors that the patient is already over-sedated.

After five propofol boluses have been given to a patient, a propofol continuous infusion will be initiated at 25mcg/kg/min. The patient may still request additional sedation with the request instrument if he or she is still conscious enough to do so. If the anesthesia provider has given more than five boluses even with the baseline propofol infusion, the infusion will be increased to 50mcg/kg/min. In the highly unlikely scenario that five additional boluses are required with a propofol infusion rate of 50 mcg/kg/min, the anesthesia providers and investigators will make a clinical decision as to what is the safest next step.

There may be scenarios that warrant conversion to general anesthesia. These scenarios include, but are not limited to, hemodynamic instability, regurgitation of gastric content, obtundation, excessive agitation, and inadequate spinal anesthesia. The decision to convert to the general anesthesia will be made by the anesthesiologist and anesthesia provider in the operating room; implementation of this study should not prevent or delay this decision if it is necessary.

Documentation will be completed by the anesthesia provider per standard protocol for electronic anesthesia charting at VCU. This will allow for data acquisition by the investigators through the anesthesiology printed record in Cerner.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing a primary elective total knee replacement by Dr. Gregory Golladay (VCU surgeon and co-investigator for this research study)
2. 18 years of age or older
3. eligible for spinal anesthesia (which will be determined by the health care providers during the standard pre-surgery clinic visits)
4. mentally capable of understanding instructions on how to request anesthesia medication
5. mentally capable of understanding instructions on how to rate pain scores, anxiety level, and patient satisfaction

Exclusion Criteria:

1. identified as a member of a regulated vulnerable population (one exception: limited English proficiency does not preclude them from this study; translation documents are available)
2. ineligibility for spinal anesthesia (which will be determined by the health care providers during the standard pre-surgery clinic visits)
3. morbid obesity, BMI greater than 40
4. allergy to propofol, midazolam, or morphine
5. pre-operative daily opioid consumption of more than 10 mg oxycodone every 6 hours
6. hearing impaired individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative propofol requirement | 2 hours
  The amount of propofol given in the operating room divided by duration of operating room time

SECONDARY OUTCOMES:
Pain score | 24 hours
  The study will collect the numerical pain scores during each four hour interval for a 24 hour time period
Satisfaction score | 72 hours
  Patient satisfaction will be determined through a hospital survey that is completed by the patient at the end of their hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Tran, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu PY, Huang ML, Lee WP, Wang C, Shih WM. Effects of music listening on anxiety and physiological responses in patients undergoing awake craniotomy. Complement Ther Med. 2017 Jun;32:56-60. doi: 10.1016/j.ctim.2017.03.007. Epub 2017 Mar 31. PMID 28619305
- [Background] Kahloul M, Mhamdi S, Nakhli MS, Sfeyhi AN, Azzaza M, Chaouch A, Naija W. Effects of music therapy under general anesthesia in patients undergoing abdominal surgery. Libyan J Med. 2017 Dec;12(1):1260886. doi: 10.1080/19932820.2017.1260886. PMID 28452603
- [Background] Li J, Zhou L, Wang Y. The effects of music intervention on burn patients during treatment procedures: a systematic review and meta-analysis of randomized controlled trials. BMC Complement Altern Med. 2017 Mar 17;17(1):158. doi: 10.1186/s12906-017-1669-4. PMID 28302117
- [Background] Alam M, Roongpisuthipong W, Kim NA, Goyal A, Swary JH, Brindise RT, Iyengar S, Pace N, West DP, Polavarapu M, Yoo S. Utility of recorded guided imagery and relaxing music in reducing patient pain and anxiety, and surgeon anxiety, during cutaneous surgical procedures: A single-blinded randomized controlled trial. J Am Acad Dermatol. 2016 Sep;75(3):585-589. doi: 10.1016/j.jaad.2016.02.1143. Epub 2016 Apr 25. PMID 27125531
- [Background] Wang Y, Tang H, Guo Q, Liu J, Liu X, Luo J, Yang W. Effects of Intravenous Patient-Controlled Sufentanil Analgesia and Music Therapy on Pain and Hemodynamics After Surgery for Lung Cancer: A Randomized Parallel Study. J Altern Complement Med. 2015 Nov;21(11):667-72. doi: 10.1089/acm.2014.0310. Epub 2015 Sep 2. PMID 26331434

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT03486106/Prot_000.pdf
  • Informed Consent Form (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT03486106/ICF_001.pdf